CLINICAL TRIAL: NCT03780322
Title: Effectiveness of Armeo Spring Pediatric in Children With Narakas I Obstetric Brachial Plexus Injury
Brief Title: Effectiveness of Armeo Spring Pediatric in Obstetric Brachial Plexus Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Pro Ayuda del Niño Lisiado (Other)
Responsible Party: Principal Investigator, Leslie Stuardo, Principal Investigator, Sociedad Pro Ayuda del Niño Lisiado
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ArmeoOBPIConcepcion
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Brachial Plexus Neuropathies; Brachial Plexus Birth Palsy
Keywords: brachial plexus birth palsy; Armeo®Spring Pediatric; physical therapy
MeSH Terms: conditions — Brachial Plexus Neuropathies | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Armeo Spring Pediatric (Experimental): This group will receive training with Armeo Spring Pediatric in 45 minute sessions, 3 times a week, for a total of 15 sessions
  Interventions: Device: Armeo Spring Pediatric
- Conventional physical and occupational therapy (Active Comparator): This group will receive combined physical and occupational therapy in 45 minute sessions, 3 times a week, for a total of 15 sessions.
  Interventions: Other: Conventional physical and occupational therapy

INTERVENTIONS:
Device: Armeo Spring Pediatric — Before intervention, the robotic device will be adjusted to the user's unique dimensions to avoid injury.
  Each 45 minute session will include active upper extremity shoulder abduction, shoulder external rotation and/or elbow extension exercises, led by virtual reality game and supported by robotic arm. Sessions will take place 3 times a week for a total of 15 sessions.
  Arms: Armeo Spring Pediatric
Other: Conventional physical and occupational therapy — Conventional therapy will combine physical and occupational therapy, including the following activities:
  1. Upper extremity weight bearing exercises.
  2. Approximation techniques on wrist, elbow and shoulder.
  3. Proprioceptive neuromuscular facilitation: shoulder flection, adduction and external rotation and shoulder flection, abduction and external rotation.
  4. Scapulothoracic joint mobilization.
  5. Stretching of shoulder abductors and external rotators.
  6. Hand/wrist facilitation exercises (with ball). This will be carried out in 45 minute sessions, 3 times a week, for a total of 15 sessions.
  Arms: Conventional physical and occupational therapy

SUMMARY:
The investigators seek to evaluate the effectiveness of Armeo®Spring Pediatric training, as compared to conventional treatment, in improving upper extremity function in children with Narakas I brachial plexus injury, aged 5-8 years, using the Mallet modified scale and passive range of movement, immediately post intervention and at 3 and 6 months´ follow up. The investigators will also monitor the appearance of adverse effects during and post intervention, with a follow up at 3 and 6 months.

DETAILED DESCRIPTION:
Obstetric brachial plexus injury is caused by damage of the cervical nerve roots C5-T1 during delivery. It has traditionally been treated with occupational and physical therapy during the first few months, evaluating at 1, 3 and 6 months if primary surgery is required. The goal of primary surgery is to repair the damaged nerve roots and restore neural function. Despite surgery, a large percentage of children will remain with varying degrees of paralysis. Since Narakas I ("Erb's") paralysis is the most common, motor sequelae usually involve limited shoulder abduction, restricted shoulder external rotation and elbow flexion contracture. This sequelae requires ongoing physical and occupational therapy, especially during school age, to ensure adequate upper extremity function and participation.

Armeo Spring Pediatric is a robotic tool that enables upper extremity training using virtual reality. Virtual reality is usually well tolerated and highly motivating to school age children. Since it's a relatively new tool, its effectiveness in the treatment of obstetric brachial plexus injury has not been documented.

This study aims to evaluate the effectiveness of Armeo Spring Pediatric training as compared to conventional therapy (occupational and physical therapy), in improving the upper extremity function of children with Narakas I (C5-C6) obstetric brachial plexus injury.

It will study two parallel groups of children ages 5-8. Both groups will receive 45 minute sessions, 3 times a week, for a total of 5 weeks (15 sessions). One group will train upper extremity function using Armeo Spring Pediatric and the other group will receive occupational and physical therapy, as detailed in protocol. They will be reevaluated at 3 and 6 months.

The appearance of adverse events, such as pain, fatigue or muscle contracture, will be documented during intervention, post intervention, and at 3 and 6 months. In the presence of one such adverse event, the training session will be suspended and the patient evaluated by physiatrist or orthopedic surgeon, with treatment if necessary. If the symptoms resolve before the next session, the patient will complete training as planned. If the symptoms are not resolved by the next session, the patient will be removed from the clinical trial until recovery.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 5 and 8 years 11 months at beginning of intervention
* Obstetric brachial plexus injury classified as Narakas I
* Legal guardian signs informed consent form

Exclusion Criteria:

* Evident shoulder or elbow dislocation during physical or radiological examination
* Elbow flexion contracture of 40º or more
* Pain during shoulder or elbow manipulation

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Change in Modified Mallet Scale | 0 weeks, 5 weeks, 17 weeks, 29 weeks
  It measures arm function in 7 different positions: arm at rest, shoulder external rotation, shoulder abduction, hand to neck, hand to mouth, hand to back and supination. Each position can be given a subscore from 1 (very altered) to 5 (almost normal), with a total score of 35. A higher score means better function (closer to normal movement or position).
  In this case, the investigators will evaluate change in Modified Mallet Scale between baseline (0 weeks), post treatment (5 weeks) and follow up (17 and 29 weeks). It will take into account changes in total scores and subscores in different positions.

SECONDARY OUTCOMES:
Upper extremity passive range of movement | 0 weeks, 5 weeks, 17 weeks and 29 weeks
  Will be measured by goniometry
Adverse events: pain. | 5 weeks, 17 weeks and 29 weeks
  Will be measured by Visual Analogue Scale. The visual analogue scale is a unidimensional measure of pain intensity. The patient marks on the line the point that they feel represents their perception of their current state. The investigator will then measure in millimeters the distance from left to right (0-100 mm) to quantify the amount of pain. A low score means less intense pain and a high score means more severe pain.
  The Visual Analogue Scale uses many formats (straight line, boxes, happy/sad faces). Because of the age of the study population in this clinical trial, the investigators have decided to use the happy/sad faces scale.
  At 5, 17 and 29 weeks, the patient will be asked to document the pain they feel at that moment, not during the treatment.
Adverse events: fatigue | 5 weeks, 17 weeks and 29 weeks
  Will be measured by Borg Scale The Borg Scale is an instrument that quantifies the exertion perceived by the patient with a score from 0-10, as follows: 0 = at rest; 1 = very easy, 2 = somewhat easy, 3 = moderate; 4 = somewhat hard, 5-6 = hard; 7-8 = really, really hard; 8-9 = really, really, really hard; 10 = maximal effort.
  At 5 weeks, the patient will be asked to document the fatigue they felt during the treatment.
  At 17 and 29 weeks, they will be asked to document the fatigue they feel at that moment.
Adverse events: muscle contracture | 5 weeks, 17 weeks and 29 weeks
  Will only be recorded if present/absent, since there is no scale to measure it

CONTACTS AND LOCATIONS:
Overall Officials: Ines Salas, MD, Study Chair — Sociedad Pro Ayuda del Niño Lisiado
Locations (1):
- Instituto Teleton, Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans-Jones G, Kay SP, Weindling AM, Cranny G, Ward A, Bradshaw A, Hernon C. Congenital brachial palsy: incidence, causes, and outcome in the United Kingdom and Republic of Ireland. Arch Dis Child Fetal Neonatal Ed. 2003 May;88(3):F185-9. doi: 10.1136/fn.88.3.f185. PMID 12719390
- [Background] Varas et al, Eventos Adversos Perinatales: Indicadores epidemiológicos, Revista Obstetricia y Ginecología 2008: 3 (2): 117-122.9
- [Background] Al-Qattan MM, El-Sayed AA, Al-Zahrani AY, Al-Mutairi SA, Al-Harbi MS, Al-Mutairi AM, Al-Kahtani FS. Narakas classification of obstetric brachial plexus palsy revisited. J Hand Surg Eur Vol. 2009 Dec;34(6):788-91. doi: 10.1177/1753193409348185. Epub 2009 Sep 28. PMID 19786407
- [Background] Vaquero G, Ramos A, Martinez JC, Valero P, Nunez-Enamorado N, Simon-De Las Heras R, Camacho-Salas A. [Obstetric brachial plexus palsy: incidence, monitoring of progress and prognostic factors]. Rev Neurol. 2017 Jul 1;65(1):19-25. Spanish. PMID 28650063
- [Background] Andersen J, Watt J, Olson J, Van Aerde J. Perinatal brachial plexus palsy. Paediatr Child Health. 2006 Feb;11(2):93-100. doi: 10.1093/pch/11.2.93. PMID 19030261
- [Background] Corkum JP, Kuta V, Tang DT, Bezuhly M. Sensory outcomes following brachial plexus birth palsy: A systematic review. J Plast Reconstr Aesthet Surg. 2017 Aug;70(8):987-995. doi: 10.1016/j.bjps.2017.05.007. Epub 2017 May 18. PMID 28602269
- [Background] El-Shamy S, Alsharif R. Effect of virtual reality versus conventional physiotherapy on upper extremity function in children with obstetric brachial plexus injury. J Musculoskelet Neuronal Interact. 2017 Dec 1;17(4):319-326. PMID 29199193
- [Background] Pellegrino G. Eficacia del tratamiento conservador en niños con parálisis braquial obstétrica. Una revisión bibliográfica. [Tesis para optar al grado de fisioterapeuta]. Tenerife España: Universidad de la Laguna; 2018. 46 p.
- [Background] Arad E, Stephens D, Curtis CG, Clarke HM. Botulinum toxin for the treatment of motor imbalance in obstetrical brachial plexus palsy. Plast Reconstr Surg. 2013 Jun;131(6):1307-1315. doi: 10.1097/PRS.0b013e31828bd487. PMID 23714792
- [Background] Yanes V, Sandobal E, Camero D, Ojeda L. Parálisis braquial obstétrica en el contexto de la rehabilitación física temprana. MediSur. 2014; 12(4): 635-649
- [Background] Gonzalez JC, Pulido JC, Fernandez F, Suarez-Mejias C. Planning, execution and monitoring of physical rehabilitation therapies with a robotic architecture. Stud Health Technol Inform. 2015;210:339-43. PMID 25991162
- [Background] Sladekova N, Kresanek J. Case report of a patient with cerebral palsy using non-robotic equipment for reeducation movements of paretic upper limb. Prz Med Uniw Rzesz Inst Leków 2014;(1):115-118
- [Background] Padyšaková H, Repková A, Sládeková N, Žiaková E, Pacek O, Musilová E, Klobucka S. Re-Education Movements of the Paretic Upper Extremity in Children age by Using Non-robotic Equipment. European Journal of Medicine 2015;8(2):106-114
- [Background] Lum PS, Burgar CG, Shor PC, Majmundar M, Van der Loos M. Robot-assisted movement training compared with conventional therapy techniques for the rehabilitation of upper-limb motor function after stroke. Arch Phys Med Rehabil. 2002 Jul;83(7):952-9. doi: 10.1053/apmr.2001.33101. PMID 12098155
- [Background] Ladenheim B, Altenburger P, Cardinal R, Monterroso L, Dierks T, Mast J, Krebs HI. The effect of random or sequential presentation of targets during robot-assisted therapy on children. NeuroRehabilitation. 2013;33(1):25-31. doi: 10.3233/NRE-130924. PMID 23949025
- [Background] You SH, Jang SH, Kim YH, Kwon YH, Barrow I, Hallett M. Cortical reorganization induced by virtual reality therapy in a child with hemiparetic cerebral palsy. Dev Med Child Neurol. 2005 Sep;47(9):628-35. PMID 16138671
- [Background] van der Sluijs JA, van Doorn-Loogman MH, Ritt MJ, Wuisman PI. Interobserver reliability of the Mallet score. J Pediatr Orthop B. 2006 Sep;15(5):324-7. doi: 10.1097/01202412-200609000-00004. PMID 16891958
- [Background] Alba-Martín, R. Fiabilidad y validez de las mediciones en hombro y codo: análisis de una aplicación de Android y un goniómetro. Rehabilitación 2016;50(2): 71-74
- [Background] Quincho, F. A., Cruz-Castillo, A. A., & Moscoso-Porras, M. G. Fiabilidad y validez de las mediciones en hombro y codo: análisis de una aplicación de Android y un goniómetro. Rehabilitación 2017; 51 (2):137
- [Background] Cole T, Robinson L, Romero L, O'Brien L. Effectiveness of interventions to improve therapy adherence in people with upper limb conditions: A systematic review. J Hand Ther. 2019 Apr-Jun;32(2):175-183.e2. doi: 10.1016/j.jht.2017.11.040. Epub 2017 Dec 29. PMID 29292028